CLINICAL TRIAL: NCT01343680
Title: A Randomized Controlled Crossover Trial of Two Different Central Venous Catheter Flushing Schemes in Pediatric Hematology and Oncology Patients in Alberta, Canada
Brief Title: Trial of Two Central Venous Catheter (CVC) Flushing Schemes in Pediatric Hematology and Oncology Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor patient accrual
Sponsor: Alberta Children's Hospital (Other)
Collaborators: Stollery Children's Hospital (Other)
Responsible Party: Principal Investigator, Martin Campbell, Paediatric Oncologist, Alberta Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ACH23736
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Childhood Cancer; Aplastic Anemia; Metabolic Disorders
MeSH Terms: conditions — Neoplasms; Anemia, Aplastic; Metabolic Diseases | interventions — Heparin; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10U/l heparin (Active Comparator)
  Interventions: Drug: Heparin
- normal saline (Experimental)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Heparin — 5ml 10 units/ml IV heparin 3 times per week
  Arms: 10U/l heparin
Drug: Normal saline — 10ml normal saline IV weekly
  Arms: normal saline

SUMMARY:
The purpose of this study is to determine whether flushing Central Venous Catheters (CVCs) with Normal saline once per week is not inferior to flushing with 10U/ml heparin 3 times per week, in preventing CVC occlusions.

DETAILED DESCRIPTION:
Tunneled central venous catheters (CVCs) are now used routinely in pediatric hematology and oncology patients. Flushing with heparin solution is routinely recommended to prevent occlusion of long term CVCs, although the concentration of heparin used, and frequency of its use varies between centres. Once weekly Normal saline is also used successfully in some pediatric enters. There is little evidence to support one method over the other.

The investigators have designed a randomised crossover trial to directly compare once weekly Normal saline flushing with 3 times per week 10U/ml heparin flushing, to determine whether Normal saline is not inferior to heparin.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of any malignant or nonmalignant disease that requires a single lumen Broviac or double lumen Hickman-type CVC for the purpose of chemotherapy, blood product support or hematopoietic stem cell transplantation.
* CVC is planned to remain in situ for 6 months from study entry

Exclusion Criteria:

* Thrombophilia (e.g. Factor V Leiden mutation, antiphospholipid syndrome) or previous thrombosis requiring anticoagulation (e.g. enoxaparin, unfractionated heparin)
* Bleeding disorder (e.g. von Willebrand's disease, hemophilia)
* Previous CVC that was removed due to any complication

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Occlusion rate | 6 months

SECONDARY OUTCOMES:
Complication rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Campbell, MBBS FRACP, Principal Investigator — Alberta Children's Hospital
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta